CLINICAL TRIAL: NCT06662877
Title: Anlotinib Plus Nab-Paclitaxels and S-1 Versus FOLFOX for Patients with Advanced Biliary Tract Cancer As Second-Line Treatment: a Phase 2/3, Multi-centric Double-stage Randomized Controlled Trial
Brief Title: Anlotinib Plus Nab-Paclitaxels and S-1 for Patients with Advanced Biliary Tract Cancer As Second-Line Treatment
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: CTTQ Pharma (Unknown)
Responsible Party: Principal Investigator, Ming Kuang, Vice President, The First Affiliated Hospital, Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2024-658
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Biliary Tract Cancer; Second Line Treatment; Chemotherapy; Tyrosine Kinase Inhibitor
Keywords: biliary tract cancer; second-line treatment; Nab-Paclitaxels; S-1; Anlotinib; FOLFOX
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Albumin-Bound Paclitaxel; tegafur-gimeracil-oteracil; S 1 (combination); anlotinib; Oxaliplatin; Leucovorin; Fluorouracil; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Experimental treatment under study
  Interventions: Drug: Albumin-bound Paclitaxel + Tegafur Gimeracil Oteracil (S-1) + Anlotinib
- Control (Active Comparator): Standard of care second-line treatment for advanced biliary tract cancer
  Interventions: Drug: Oxaliplatin + Leucovorin + Fluorouracil (FOLFOX regimen)

INTERVENTIONS:
Drug: Albumin-bound Paclitaxel + Tegafur Gimeracil Oteracil (S-1) + Anlotinib — Albumin-bound Paclitaxel, 125mg/m2,iv.drip,d1,d8,Q3W +Tegafur Gimeracil Oteracil (S-1) 40-60mg,p.o,bid,d1-d14,Q3W+Anlotinib 10mg,p.o,d1-d14,Q3W
  Arms: Experimental
Drug: Oxaliplatin + Leucovorin + Fluorouracil (FOLFOX regimen) — Oxaliplatin 85 mg/m2,d1,iv.drip,Q2W + Leucovorin 400mg/m2,d1,iv.drip,Q2W+ Fluorouracil 2400 mg/m2 civ46h, Q2W
  Arms: Control

SUMMARY:
Biliary tract cancer (BTC) presents with a 5-year survival rate less than 5%. The goal of this clinical trial is to evaluate if Anlotinib plus Nab-Paclitaxels and S-1 as second-line regimen can improve the treatment efficacy in advanced biliary tract cancer (BTC) after progression upon first-line standard treatment, in comparison with standard second-line FOLFOX regimen.

DETAILED DESCRIPTION:
Biliary tract cancer (BTC) mainly includes intrahepatic cholangiocarcinoma, hilar cholangiocarcinoma, extrahepatic cholangiocarcinoma and gallbladder carcinoma, and the 5-year survival rate is less than 5%. Most patients were diagnosed as advanced stage, and missed the opportunity of radical surgery. ABC-02 study established gemcitabine combined with platinum drugs as the first-line standard treatment for unresectable BTC. However, after the disease progresses, the second-line treatment options and efficacies are limited. In recent years, BTC second-line treatment has made some breakthroughs in the field of chemotherapy and targeted therapy. However, the benefits of chemotherapy, immunotherapy and targeted drugs alone in the second line treatment of BTC is unsatisfactory. The combined scheme of two or three drugs sees the possibility of patients benefiting, but it still needs better scheme design and larger sample size for further verification. A phase II single-arm small-sample clinical trial exploring albumin-bound paclitaxel combined with S-1 capsule in the first-line treatment of advanced biliary adenocarcinoma initially showed the efficacy and safety of AS regimen in cholangiocarcinoma, and the efficacy and safety of Anlotinib in BTC were also confirmed in the small-sample study. Therefore, this study intends to explore the efficacy and safety of the second-line treatment of advanced BTC with Anlotinib combined with AS chemotherapy in comparison with the establised standard second-line regimen (FOLFOX).

ELIGIBILITY:
Inclusion Criteria:

1. Signed a written informed consent form before enrollment;
2. Age >18 years, both male and female are eligible;
3. Patients with pathologically confirmed advanced biliary tract that has progressed after first-line gemcitabine-based therapy;
4. Have measurable lesions (according to RECIST 1.1 criteria, non-lymph node lesions with a long diameter ≥10 mm on CT scan, or lymph node lesions with a short diameter ≥15 mm on CT scan);
5. ECOG Performance Status (PS) score: 0-1;
6. Expected survival time longer than 12 weeks;
7. Key organ functions meet the following criteria (without the use of any blood components or growth factors within 14 days): Hematology: Neutrophils ≥1.5×10⁹/L; Platelet count ≥100×10⁹/L; Hemoglobin ≥ 90 g/L; Liver and kidney function: Serum creatinine (SCr) ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance rate ≥50 ml/min (Cockcroft-Gault formula); Total bilirubin (TBIL) ≤ 1.5 times the ULN; Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels ≤ 2.5 times the ULN (if abnormal liver function is due to liver metastasis, then ≤ 5 times the ULN); urine protein < 2+; if urine protein ≥ 2+, 24-hour urine protein quantification must show protein ≤1g;
8. Normal coagulation function, no active bleeding or thrombotic diseases: International Normalized Ratio (INR) ≤ 1.5 × ULN; Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN; Prothrombin Time (PT) ≤ 1.5 × ULN;
9. The subject voluntarily participates in this study, has good compliance, and is willing to cooperate with safety and survival follow-ups.

Exclusion Criteria:

1. Subjects with a history of or concurrent malignancies, except for cured basal cell carcinoma of the skin or carcinoma in situ of the cervix;
2. Known allergy to macromolecular protein preparations or known hypersensitivity to the components of the administered drugs;
3. Subjects with existing thyroid dysfunction that cannot be maintained within the normal range by medication;
4. Uncontrolled hypertension despite optimal treatment, defined as systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg;
5. Subjects with uncontrolled cardiac clinical symptoms or diseases, such as: (1) heart failure above NYHA class II, (2) unstable angina, (3) myocardial infarction within the past year, (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
6. Subjects with any active autoimmune disease or a history of autoimmune disease;
7. Subjects using immunosuppressive agents or systemic or absorbable local corticosteroids for immunosuppressive purposes (prednisone dose >10 mg/day or equivalent efficacy corticosteroids) who continue to use them within 2 weeks before enrollment;
8. Subjects with central nervous system metastases;
9. Subjects with active infections or unexplained fever >38.5°C during screening or before the first dose (subjects with tumor-related fever, as judged by the investigator, may be enrolled);
10. Subjects with significant hemoptysis (fresh blood) within 2 months before enrollment or daily hemoptysis volume ≥2.5 ml;
11. Subjects with any condition that may increase the risk of gastrointestinal bleeding or perforation, such as active peptic ulcers, known intraluminal metastatic lesions, inflammatory bowel disease, history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days before the start of the study;
12. Subjects with a history or current evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis, or severely impaired lung function;
13. Subjects with a history or current evidence of bronchiectasis, cavitary pulmonary tuberculosis, lung abscess, rheumatic heart disease with mitral valve stenosis, or cardiogenic pulmonary edema, which could cause hemoptysis;
14. Subjects with congenital or acquired immune deficiencies, such as those infected with HIV or with active hepatitis (transaminase levels not meeting inclusion criteria, hepatitis B reference: HBV DNA ≥1000 IU/ml; hepatitis C reference: HCV RNA ≥1000 IU/ml);
15. Subjects who have received or may receive a live vaccine within 4 weeks before or during the study;
16. Subjects with a known history of psychiatric drug abuse, alcoholism, or drug addiction;
17. Pregnant or breastfeeding women or those planning to conceive during the study period;
18. Subjects whom the investigator deems should be excluded from the study, such as those with factors that may lead to early termination of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2024-11-25 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From randomisation to death, up to 5 years
  Overall Survival (OS), defined as the time between the date of the subject's first dose and the subject's death from all causes. The OS of subjects who were alive at the time of the final follow-up visit was counted as data censored at the time of the final follow-up visit.
Progression-Free Survival | From randomisation to disease progression or death, up to 5 years
  Progression-Free Survival (PFS) is defined as the time from the date of the subject's first dose of medication to the date of the first documented tumor progression (assessed according toRECIST 1.1 criteria, with or without continuation of treatment) or the date of death from anycause, whichever occurs first. The median PFS and its 95% Cl will be analyzed using the Kaplan-Meier method and survival graphs will be plotted.

SECONDARY OUTCOMES:
Objective Response Rate | From randomisation, up to 5 years
  Refers to the proportion of patients whose tumors shrank by a certain amount and remained sofor a certain period of time, and includes both CR and PR cases. Objective tumor remission was assessed using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criteria).
Disease control rate | From randomisation, up to 5 years
  Refers to the proportion of patients whose tumors shrank by a certain amount and remained sofor a certain period of time, and includes both CR and PR cases. Obiective tumor remission was assessed using the Solid Tumor Remission Assessment Criteria (RECIST 1.1 criterial

OTHER OUTCOMES:
Quality of Life | From baseline, every 3weeks until end of treatment, an average of 4-6 months
  Patients' quality of life was assessed according to the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30), assessed at baseline and every 3 weeks thereafter
Adverse Events | From randomisation, up to 5 years
  Defined as the proportion of grade ≥3 hematologic or non-hematologic toxic events occurring from the start of medication to the end of follow-up. Adverse events include, but are not limited to, liver dysfunction, hematologic system damage, pulmonary toxicity, and ocular toxicity. The severity of adverse events will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE v5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang W, Sun Y, Jiang Z, Qu W, Gong C, Zhou A. Nab-paclitaxel plus tegafur gimeracil oteracil potassium capsule (S-1) as first-line treatment for advanced biliary tract adenocarcinoma: a phase 2 clinical trial. Hepatobiliary Surg Nutr. 2023 Feb 28;12(1):37-44. doi: 10.21037/hbsn-21-172. Epub 2021 Oct 18. PMID 36860259
- [Background] Shen G, Zheng F, Ren D, Du F, Dong Q, Wang Z, Zhao F, Ahmad R, Zhao J. Anlotinib: a novel multi-targeting tyrosine kinase inhibitor in clinical development. J Hematol Oncol. 2018 Sep 19;11(1):120. doi: 10.1186/s13045-018-0664-7. PMID 30231931
- [Background] Klein O, Kee D, Nagrial A, Markman B, Underhill C, Michael M, Jackett L, Lum C, Behren A, Palmer J, Tebbutt NC, Carlino MS, Cebon J. Evaluation of Combination Nivolumab and Ipilimumab Immunotherapy in Patients With Advanced Biliary Tract Cancers: Subgroup Analysis of a Phase 2 Nonrandomized Clinical Trial. JAMA Oncol. 2020 Sep 1;6(9):1405-1409. doi: 10.1001/jamaoncol.2020.2814. PMID 32729929
- [Background] Li X, Zhou N, Yang Y, Lu Z, Gou H. Efficacy and biomarker analysis of second-line nab-paclitaxel plus sintilimab in patients with advanced biliary tract cancer. Cancer Sci. 2024 Jul;115(7):2371-2383. doi: 10.1111/cas.16179. Epub 2024 Apr 18. PMID 38638055
- [Background] Lim SH, Hong JY, Park JO, Park YS, Kim ST. Pemetrexed and Erlotinib as a Salvage Treatment in Patients With Metastatic Biliary Tract Cancer Who Failed Gemcitabine-containing Chemotherapy: A Phase II Single-arm Prospective Study. Anticancer Res. 2023 Sep;43(9):4161-4167. doi: 10.21873/anticanres.16607. PMID 37648323
- [Background] Abou-Alfa GK, Macarulla T, Javle MM, Kelley RK, Lubner SJ, Adeva J, Cleary JM, Catenacci DV, Borad MJ, Bridgewater J, Harris WP, Murphy AG, Oh DY, Whisenant J, Lowery MA, Goyal L, Shroff RT, El-Khoueiry AB, Fan B, Wu B, Chamberlain CX, Jiang L, Gliser C, Pandya SS, Valle JW, Zhu AX. Ivosidenib in IDH1-mutant, chemotherapy-refractory cholangiocarcinoma (ClarIDHy): a multicentre, randomised, double-blind, placebo-controlled, phase 3 study. Lancet Oncol. 2020 Jun;21(6):796-807. doi: 10.1016/S1470-2045(20)30157-1. Epub 2020 May 13. PMID 32416072
- [Background] Merters J, Lamarca A. Integrating cytotoxic, targeted and immune therapies for cholangiocarcinoma. J Hepatol. 2023 Mar;78(3):652-657. doi: 10.1016/j.jhep.2022.11.005. Epub 2022 Nov 15. PMID 36400328
- [Background] Yoo C, Kim KP, Jeong JH, Kim I, Kang MJ, Cheon J, Kang BW, Ryu H, Lee JS, Kim KW, Abou-Alfa GK, Ryoo BY. Liposomal irinotecan plus fluorouracil and leucovorin versus fluorouracil and leucovorin for metastatic biliary tract cancer after progression on gemcitabine plus cisplatin (NIFTY): a multicentre, open-label, randomised, phase 2b study. Lancet Oncol. 2021 Nov;22(11):1560-1572. doi: 10.1016/S1470-2045(21)00486-1. Epub 2021 Oct 14. PMID 34656226
- [Background] Lamarca A, Palmer DH, Wasan HS, Ross PJ, Ma YT, Arora A, Falk S, Gillmore R, Wadsley J, Patel K, Anthoney A, Maraveyas A, Iveson T, Waters JS, Hobbs C, Barber S, Ryder WD, Ramage J, Davies LM, Bridgewater JA, Valle JW; Advanced Biliary Cancer Working Group. Second-line FOLFOX chemotherapy versus active symptom control for advanced biliary tract cancer (ABC-06): a phase 3, open-label, randomised, controlled trial. Lancet Oncol. 2021 May;22(5):690-701. doi: 10.1016/S1470-2045(21)00027-9. Epub 2021 Mar 30. PMID 33798493
- [Background] Lamarca A, Hubner RA, David Ryder W, Valle JW. Second-line chemotherapy in advanced biliary cancer: a systematic review. Ann Oncol. 2014 Dec;25(12):2328-2338. doi: 10.1093/annonc/mdu162. Epub 2014 Apr 25. PMID 24769639
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Background] Ilyas SI, Affo S, Goyal L, Lamarca A, Sapisochin G, Yang JD, Gores GJ. Cholangiocarcinoma - novel biological insights and therapeutic strategies. Nat Rev Clin Oncol. 2023 Jul;20(7):470-486. doi: 10.1038/s41571-023-00770-1. Epub 2023 May 15. PMID 37188899